CLINICAL TRIAL: NCT01848925
Title: A Phase I Open-label, Randomized, Safety and Efficacy Study of SANGUINATE™ at Two Doses Levels Versus Hydroxyurea in Sickle Cell Disease (SCD) Patients.
Brief Title: Study of SANGUINATE™ Versus Hydroxyurea in Sickle Cell Disease (SCD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGSC-003
Record Dates: First submitted 2013-04-23; First posted 2013-05-08 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Sickle Cell Disease
Keywords: SANGUINATE
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — PEGylated carboxyhemoglobin bovine; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SANGUINATE™ (Experimental): PEG-bHb-CO
  Interventions: Biological: SANGUINATE™
- Hydroxyurea (Active Comparator): Standard of care for Sickle Cell treatment, 15 mg/kg.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Biological: SANGUINATE™ — 40 mg/mL intravenous infusion.
  Arms: SANGUINATE™
Drug: Hydroxyurea — Standard of care for Sickle Cell treatment, 15 mg/kg.
  Other Names: Hydroxycarbamide; Brand Names includes: Hydria, Droxia.
  Arms: Hydroxyurea

SUMMARY:
The purpose of this study is to compare the safety of SANGUINATE™ versus Hydroxyurea in patients suffering from Sickle Cell Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Homozygous (HbSS) Sickle Cell Anemia;
* Hb levels: >6g/dL - <10g/dL;
* Age : >18 years old;
* Frequency of ER hospitalizations < 6x/yr for SCD pain events documented "medical history".

Exclusion Criteria:

* Patients, who are on chronic transfusion program, defined as regular transfusions every 2-8 weeks;
* Allergic to Hydroxyurea;
* History of clinical significant disease, as determined by the Investigator;
* History of allergy or major allergic reaction considered to be clinically significant by the Investigator;
* Screening assessments considered to be abnormal by the Investigator;
* Patient has sever pulmonary hypertension (index >3 meters per sec);
* Donated blood within 60 days of screening or otherwise experienced blood loss of >250 mL within the same period;
* Intending to begin new concomitant drug therapy or over-the-counter medication anytime from scree4nin to the time of administration of study drug;

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To Compare SANGUINATE™ and Hydroxyurea in Sickle Cell Disease patients. | 7 days
  Compare pain management between SANGUINATE™ and Hydroxyurea using 0-10 Numeric Pain Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kenny M Galvez, MD, Principal Investigator — Hospital Pablo Tobin Uribe; Luis F Uribe, MD, Principal Investigator — Fundacion Reina Isabel; Nestor Sosa, MD, Principal Investigator — Hospital Punta Pacifica; Angel Hernandez, MD, Principal Investigator — Fundacion BIOS
Locations (4):
- Colombia (3):
  - Fundacion BIOS, Barranquilla
  - Fundacion Reina Isabel, Cali
  - Hospital Pablo TobinUribe, Medellín
- PAMRI, Panama City, Panama